CLINICAL TRIAL: NCT02457715
Title: Feasibility of a Consumer Based Accelerometer in Monitoring Outpatient Physical Activity: A Study in Patients With Cancer and Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00063108
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer; Renal Cancer; Brain Cancer; ALS
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prostate Cancer: Subjects will use a Jawbone Up24 for 14 weeks.
- Renal Cancer: Subjects will use a Jawbone Up24 for 14 weeks.
- Brain Cancer: Subjects will use a Jawbone Up24 for 14 weeks.
- Amyotrophic Lateral Sclerosis (ALS): Subjects will use a Jawbone Up24 for 14 weeks.

SUMMARY:
This is a parallel group, single institution, prospective clinical study. The purpose of this study is to assess whether the Jawbone Up 24, a consumer based accelerometer, can be a feasible tool to study physical activity in cancer patients and patients with Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Patients > = 18 years of age.
* Patient must be able to ambulate and complete the 6 minute walk test without use of a walker, cane, or any assist devices.
* Cancer patients or ALS patients who meet the following criteria:

Prostate cancer:

* Histologically confirmed prostate cancer.
* Patients who are initiating any chemotherarpy (examples are docetaxel, cabazitaxel, etc.) and/or hormone directed treatment for prostate cancer. Examples of hormone directed therapy include GnRH agonist or antagonists (such as leuprolide, goserelin, triptorelin, histrelin and degarelix), androgen receptor blockers (such as bicalutamide or enzalutamide), or androgen biosynthesis inhibitors (such as abiraterone).

Renal cancer:

* Histologically confirmed renal cell carcinoma (RCC).
* Metastatic disease, in the opinion of the treating provider.
* Starting any systemic therapy for metastatic disease

Brain cancer:

* Histologically confirmed high grade glioma.
* Status post concurrent radiation therapy and daily temozolomide.
* Starting adjuvant temozolomide therapy.

ALS patients who are:

* Already on a stable dose of Riluzole for at least one month.
* ALSFRS-R with <or equal to 2 point decline in last month.
* Must have ALSFRS-R walking score of at least 3 or 4 and FVC at least 50% (to ensure patients are fit enough for ambulation and physical activity).

  - Technology requirement:
* Patients will need to own a smart phone that can interface with the Jawbone Up 24.
* Patients willing to provide their own internet access for this study. This will include either a data plan or Wi-Fi access on the patient's smart phone for use of the Jawbone App. They will also need internet access (through their smart phone or home computer) for setting up a SGHIx account. Patients are welcome to use the free guest Wi-Fi access within the Duke Outpatient clinic area for the purpose of this study.
* Patients will need a home computer or adaptor with USB port to charge the Jawbone Up 24.

Exclusion Criteria:

* Non-English Speaking or inability to read and understand English
* Presence of cardiovascular disease that would make physical activity risky at the discretion of the provider.
* Any patient who is unable to comprehend and operate the activity tracker at the discretion of the enrolling provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a parallel group, single institution, prospective clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Compliance rate of cancer and ALS patients using the device during a 14 week period. | 14 weeks

SECONDARY OUTCOMES:
Number of steps per day in cancer patients. | 14 weeks
Karnofsky performance status in cancer patients. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States